CLINICAL TRIAL: NCT00261235
Title: A Randomized Trial of Supported Employment Versus USES Enhanced Supported Employment in Veterans With Serious Mental Illness
Brief Title: Trial of Supported Employment Versus USES Supported Employment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sandra Resnick, Principal Investigator, VA Connecticut Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SR0007; MIRECC
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Mental Disorders
Keywords: Rehabilitation, Vocational; Virtues; Employment, supported; veterans; Mentally Ill Persons
MeSH Terms: conditions — Mental Disorders | interventions — Employment, Supported

INTERVENTIONS:
Behavioral: Supported Employment
Behavioral: Using Strengths in Employment System (USES)

SUMMARY:
The purpose of this study is to test the effectiveness of USES, a strengths-based enhancement to supported employment (SE), as compared to supported employment alone.

DETAILED DESCRIPTION:
The objective of this study is to test the effectiveness of supported employment plus Using Strengths in Employment Services (USES), an enhancement to supported employment that seeks to identify and increase the use of personal strengths, as compared to supported employment alone, for veterans with severe mental illness and/or substance abuse disorders. We hypothesize that rates of competitive employment will be greater in the experimental group than the control group. We also expect that individuals in the USES group will have greater job tenure, and will show greater improvements in recovery measures such as empowerment, self-efficacy and self-esteem.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Unemployed
* Referred by clinician to SE services
* Able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-03; Primary Completion 2006-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
job tenure (cumulative throughout course of study)

SECONDARY OUTCOMES:
empowerment
self-efficacy
self-esteem

CONTACTS AND LOCATIONS:
Overall Officials: Sandra G. Resnick, Ph.D., Principal Investigator — VA Northeast Program Evaluation Center
Locations (2):
- United States (2):
  - West Haven VAMC, West Haven, Connecticut
  - Syracuse VA Healthcare System, Syracuse, New York